CLINICAL TRIAL: NCT04656977
Title: Évaluer l'efficacité d'Une Intervention en réalité Virtuelle Sur le Bien-être Des Femmes Ayant vécu un décès périnatal : un Essai contrôlé randomisé
Brief Title: Providing Psychological and Emotional Support After Perinatal Loss: A Virtual Reality-Based Intervention
Acronym: DIANE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universite du Quebec en Outaouais (Other)
Collaborators: Canadian Research Chair in Family Psychosocial Health (Unknown); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Giulia Corno, Postdoctoral fellow, Universite du Quebec en Outaouais
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-867
Record Dates: First submitted 2020-11-10; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Grief; Perinatal
Keywords: Perinatal loss; Perinatal grief; Women mental health; Virtual reality; Psychological intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR+TAU (Active Comparator): Participants will participate first to a VR-based intervention and then to the TAU condition. The TAU condition is a homogenous standard program proposed by the Centre d'études et de recherché en intervention familiale (CERIF) at Université du Québec en Outaouais (UQO) based on group counseling offered to women and men who experienced a perinatal loss.
  Interventions: Other: VR; Other: TAU
- TAU+VR (Active Comparator): Participants will be invited first to participate to the TAU condition and then to the VR-based intervention.
  Interventions: Other: VR; Other: TAU

INTERVENTIONS:
Other: VR — The proposed intervention will consist in three weekly sessions of 2h focused, respectively, on: (1) gathering information about the loss and psychoeducation about perinatal grief, and introduction to the virtual environment; (2) through the use of the virtual environment, women will be assisted in the elaboration and acceptation of loss; (3) recreate, using the features of the virtual environment (i.e., a series of different virtual landscapes and symbolic elements personalized to each participant as personal pictures, sounds or videos) a new and positive metaphor representing the woman's future life.
  Other Names: VR-based intervention
Other: TAU — The TAU condition is a homogenous standard program proposed by the CERIF at UQO based on group counseling offered to women and men who experienced a perinatal loss.
  Other Names: Group counseling

SUMMARY:
The loss of an infant during the perinatal period has been recognized as a complex and potentially traumatic life event and can have a significant impact on women's mental health. However, often times, psychological aftercare is typically not offered, and manualized interventions are rarely used in clinical care practice and have seldom been evaluated. In recent years, a growing number of studies have demonstrated the efficacy of virtual reality (VR) interventions to facilitate the expression and coping with emotions linked to a traumatic event. The objective of the proposed paper is to present the protocol of a randomized control trial aimed to assess a novel VR-based intervention for mothers who experienced a perinatal loss. The investigators hypothesize that the VR-based intervention group will show significantly reduced symptoms related to grief, postnatal depression and general psychopathology after treatment relative to a treatment-as-usual (TAU) group. With the present study the investigators propose to answer to the unquestionable need for interventions addressed to ameliorate the emotional effects in women who experienced perinatal loss, by exploiting also the therapeutic opportunities offered by a new technology as VR.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who had recently experienced a perinatal death, including: having lost a child during pregnancy because of miscarriage (i.e., embryo or fetus death prior the 28th week of gestation); termination due to medical indications; stillbirth (i.e., fetus death after 28 completed weeks of gestation); or neonatal death (i.e., infant death within the first 7 days of life).
* Women who have experienced perinatal death while pregnant within no more than 1 year before the enrollment will be invited to participate to the study.

Exclusion Criteria:

* Significant vision impairments despite wearing corrective glasses or lenses.
* Presence of a severe and disabling diagnosed mental disorder which requires immediate treatment.
* Being under psychological treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Perinatal Grief Scale (change) | Day 1 (pre-assessment), up to 3 weeks from day 1, up to 6 weeks from day 1
Inventory of Complicated Grief (change) | Day 1 (pre-assessment), up to 3 weeks from day 1, up to 6 weeks from day 1
Beck Depression Inventory-II (change) | Day 1 (pre-assessment), up to 3 weeks from day 1, up to 6 weeks from day 1
Edinburgh Postnatal Depression Scale (change) | Day 1 (pre-assessment), up to 3 weeks from day 1, up to 6 weeks from day 1
State and Trait Anxiety Inventory form Y (change) | Day 1 (pre-assessment), up to 3 weeks from day 1, up to 6 weeks from day 1
Positive and Negative Affect Scale (change) | Day 1 (pre-assessment), up to 3 weeks from day 1, up to 6 weeks from day 1
Clinical Global Impression rated by the therapist (change) | Day 1 (pre-assessment), up to 3 weeks from day 1, up to 6 weeks from day 1

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire | Up to 3 weeks from day 1, up to 6 weeks from day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Université du Québec en Outaouais, Gatineau, Quebec, Canada

REFERENCES:
- [Background] Corno G, Bouchard S, Banos RM, Rivard MC, Verdon C, de Montigny F. Providing Psychological and Emotional Support After Perinatal Loss: Protocol for a Virtual Reality-Based Intervention. Front Psychol. 2020 Jun 10;11:1262. doi: 10.3389/fpsyg.2020.01262. eCollection 2020. PMID 32587557